CLINICAL TRIAL: NCT06132321
Title: Monocentric Prospective Observational Multiparametric Study on the Quality of Life in Patients Undergone Surgery for Vulvar Cancer and Reconstruction (3233)
Brief Title: Quality of Life in Patients Undergone Vulvar Reconstruction After Vulvar Cancer Resection (3233)
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Gentileschi Stefano, Associate Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3233
Record Dates: First submitted 2023-03-11; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Vulvar Neoplasms
Keywords: Vulvar Neoplasms; Vulvar cancer; Vulvar Reconstruction; Vulvoperineal Reconstruction; Gynecological Cancer; Quality of Life
MeSH Terms: conditions — Vulvar Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients operated for vulvar cancer without reconstruction
  Interventions: Behavioral: Quality of life questionnaires
- Patients operated for vulvar cancer with reconstruction
  Interventions: Behavioral: Quality of life questionnaires

INTERVENTIONS:
Behavioral: Quality of life questionnaires — Detecting by mean of questionnaires quality of life, urinary function, pain, sexual function and lymphedema status before and after surgery for vulvar cancer, associated or not to vulvar reconstruction

SUMMARY:
This study aims to evaluate the patients'quality of life before and after surgery for vulvar cancer and reconstruction, employing different questionnaires and investigating different items.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery for vulvar cancer
* Patients providing consent to be enrolled in the study

Exclusion Criteria:

* Cognitive impairment
* psychiatric disorder
* neurodegenerative disorder

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing ablative surgery for vulvar cancer associated or not to vulvoperineal reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 93 (Estimated)
Dates: Start 2020-06-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rand 36 | June 2020 - June 2025
  Changes in RAND-36 score before and after surgery

SECONDARY OUTCOMES:
ICIQ-SF | June 2020 - June 2025
  Changes in ICIQ-SF score before and after surgery
FSFI | June 2020 - June 2025
  Changes in FSFI score before and after surgery
ECOG | June 2020 - June 2025
  Changes in ECOG score before and after surgery
LYM-LEG-QoL | June 2020 - June 2025
  Changes in LYM-LEG-QoL score before and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Gentileschi, Prof., Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2013. CA Cancer J Clin. 2013 Jan;63(1):11-30. doi: 10.3322/caac.21166. Epub 2013 Jan 17. PMID 23335087
- [Result] Rajaram S, Gupta B. Management of Vulvar Cancer. Rev Recent Clin Trials. 2015;10(4):282-8. doi: 10.2174/1574887110666150923112723. PMID 26411953
- [Result] Hellinga J, Te Grootenhuis NC, Werker PMN, de Bock GH, van der Zee AGJ, Oonk MHM, Stenekes MW. Quality of Life and Sexual Functioning After Vulvar Reconstruction With the Lotus Petal Flap. Int J Gynecol Cancer. 2018 Nov;28(9):1728-1736. doi: 10.1097/IGC.0000000000001340. PMID 30157166
- [Result] Dessole M, Petrillo M, Lucidi A, Naldini A, Rossi M, De Iaco P, Marnitz S, Sehouli J, Scambia G, Chiantera V. Quality of Life in Women After Pelvic Exenteration for Gynecological Malignancies: A Multicentric Study. Int J Gynecol Cancer. 2018 Feb;28(2):267-273. doi: 10.1097/IGC.0000000000000612. PMID 26807639
- [Result] Froeding LP, Greimel E, Lanceley A, Oberguggenberger A, Schmalz C, Radisic VB, Nordin A, Galalaei R, Kuljanic K, Vistad I, Schnack TH, Jensen PT; European Organization of Research Treatment of Cancer Quality of Life Group the Gynecological Cancer group. Assessing Patient-reported Quality of Life Outcomes in Vulva Cancer Patients: A Systematic Literature Review. Int J Gynecol Cancer. 2018 May;28(4):808-817. doi: 10.1097/IGC.0000000000001211. PMID 29420364
- [Result] Saimanen I, Kuosmanen V, Rahkola D, Selander T, Karkkainen J, Harju J, Aspinen S, Eskelinen M. RAND-36-Item Health Survey: A Comprehensive Test for Long-term Outcome and Health Status Following Surgery. Anticancer Res. 2019 Jun;39(6):2927-2933. doi: 10.21873/anticanres.13422. PMID 31177131
- [Result] Gentileschi S, Servillo M, Garganese G, Fragomeni S, De Bonis F, Scambia G, Salgarello M. Surgical therapy of vulvar cancer: how to choose the correct reconstruction? J Gynecol Oncol. 2016 Nov;27(6):e60. doi: 10.3802/jgo.2016.27.e60. Epub 2016 Jul 12. PMID 27550406
- [Result] Gentileschi S, Caretto AA, Servillo M, Stefanizzi G, Alberti C, Garganese G, Fragomeni SM, Federico A, Tagliaferri L, Moroni R, Scambia G. Feasibility, indications and complications of SCIP flap for reconstruction after extirpative surgery for vulvar cancer. J Plast Reconstr Aesthet Surg. 2022 Mar;75(3):1150-1157. doi: 10.1016/j.bjps.2021.11.005. Epub 2021 Nov 13. PMID 34866009
- [Result] Caretto AA, Stefanizzi G, Fragomeni SM, Federico A, Tagliaferri L, Lancellotta V, Scambia G, Gentileschi S. Lymphatic Function of the Lower Limb after Groin Dissection for Vulvar Cancer and Reconstruction with Lymphatic SCIP Flap. Cancers (Basel). 2022 Feb 21;14(4):1076. doi: 10.3390/cancers14041076. PMID 35205824